CLINICAL TRIAL: NCT02296866
Title: Assessment of Prokinetic Effects of Erythromycin in Emergency Patients With a Full Stomach
Status: Completed | Type: Observational
Sponsor: Lionel Bouvet (Other)
Responsible Party: Sponsor-Investigator, Lionel Bouvet, MD PhD, Hôpital Edouard Herriot
Organization: Hôpital Edouard Herriot (Other)
Other Study IDs: 2013-A01257-38
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Emergency Surgery; Full Stomach

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The aims of the study is to assess whether the intravenous infusion of 3 mg/kg erythromycin has a significant gastrokinetic effect leading to empty the stomach in less than 90 minutes in non-fasting patients undergoing emergency trauma surgery.

ELIGIBILITY:
Inclusion Criteria:

* Emergency surgery for trauma
* ASA 1 and 2 patients
* Full stomach (antral area > 550 mm²)
* Adult patients

Exclusion Criteria:

* No contraindication to erythromycin
* Extreme emergency surgery (time frame < 90 min between arrival in the service and the start of the surgery)
* gastroparesis or pathology associated with gastroparesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all trauma patients with a full stomach, undegoing emergency surgery
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
ultrasonographic measurement of antral area | 30 minutes and immediately before erythromycin infusion, and 30, 60 and 90 min after the start of erythromycin infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Edouard Herriot, Lyon, France